CLINICAL TRIAL: NCT05165771
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2 Proof-of-Concept Study to Evaluate Safety, Tolerability, and Efficacy of GS-5718 on Background Therapy With Conventional Synthetic Disease-modifying Antirheumatic Drug(s) (csDMARDs) in Participants With Active Rheumatoid Arthritis Who Have an Inadequate Response to Biologic DMARD(s) Treatment
Brief Title: Study to Evaluate Safety, Tolerability, and Efficacy of GS-5718 in Participants With Active Rheumatoid Arthritis Who Have an Inadequate Response to Disease-modifying Antirheumatic Drug(s) (bDMARDs) Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to withdraw study.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-561-5898; 2021-002664-52 (EudraCT Number)
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GS-5718 Dose A (Experimental): Participants will receive GS-5718 Dose A once daily + placebo to match (PTM) GS-5718 Dose B once daily + PTM tofacitinib twice daily for up to 12 weeks.
  Interventions: Drug: GS-5718; Drug: Placebo to match GS-5718; Drug: Placebo to match Tofacitinib
- GS-5718 Dose B (Experimental): Participants will receive GS-5718 Dose B once daily + PTM GS-5718 Dose A once daily + PTM tofacitinib twice daily for up to 12 weeks.
  Interventions: Drug: GS-5718; Drug: Placebo to match GS-5718; Drug: Placebo to match Tofacitinib
- Tofacitinib (Active Comparator): Participants will receive tofacitinib 5 mg twice daily + PTM GS-5718 (Dose A + Dose B) once daily for up to 12 weeks.
  Interventions: Drug: Placebo to match GS-5718; Drug: Tofacitinib 5 mg
- Placebo (Placebo Comparator): Participants will receive PTM GS-5718 (Dose A + Dose B) once daily + PTM tofacitinib twice daily for up to 12 weeks.
  Interventions: Drug: Placebo to match GS-5718; Drug: Placebo to match Tofacitinib

INTERVENTIONS:
Drug: GS-5718 — Tablets administered orally
  Arms: GS-5718 Dose A
Drug: GS-5718 — Tablets administered orally
  Arms: GS-5718 Dose B
Drug: Placebo to match GS-5718 — Tablets administered orally
Drug: Tofacitinib 5 mg — Tablets administered orally
  Other Names: XELJANZ®
  Arms: Tofacitinib
Drug: Placebo to match Tofacitinib — Tablets administered orally
  Arms: GS-5718 Dose A; GS-5718 Dose B; Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of GS-5718 versus placebo for the treatment of rheumatoid arthritis (RA) as measured by change from baseline in Disease Activity Score (DAS) based on 28 joints using C-reactive protein (CRP) (DAS28[CRP]) at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) ≥ 3 months prior to screening fulfilling the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA
* Rheumatoid factor (RF) and/or anti-citrullinated protein antibodies (ACPA) positivity
* Individual fulfills all of the following minimum disease activity criteria:

  * ≥ 6 swollen joints (from a swollen joint count based on 66 joints [SJC66]) provided this would also fulfill ≥ 4 swollen joints (from a swollen joint count based on 28 joints [SJC28]) at screening and Day 1, and
  * ≥ 6 tender joints (from a tender joint count based on 68 joints [TJC68]), provided this would also fulfill ≥ 4 tender joints (from a tender joint count based on 28 joints [TJC28]) at screening and Day 1, and
  * hsCRP > upper limit of normal at screening
* Received at least one bDMARD for the treatment of RA to which there is a lack of efficacy and/or intolerance.

Key Exclusion Criteria:

* Individuals who do not qualify per the tofacitinib label and/or local guidelines should not be enrolled.
* Prior exposure to any Janus kinase inhibitor

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Disease Activity Score (DAS) Based on 28 Joints Using C-reactive Protein (CRP) DAS28 (CRP) at Week 12 | Baseline, Week 12
  The DAS28(CRP) is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), subject's global assessment (SGA) of disease activity assessed using visual analog scale (VAS) on a scale of 0-100 (0 indicating no arthritis and 100 indicating extremely active arthritis), and high-sensitivity C-reactive protein (hsCRP) measurement for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve American College of Rheumatology 20% Improvement (ACR20) Response at Week 12 | Week 12
  ACR20 response is achieved when the participant has: ≥20% improvement (reduction) from baseline in tender joint count based on 68 joints (TJC68), swollen joint count based on 66 joints (SJC66) and in at least 3 of the following 5 items: physician's global assessment of disease activity (PGA) assessed using VAS on a scale of 0-100 (0 indicating no disease activity and 100 indicating maximum disease activity) and SGA assessed using VAS on a scale of 0-100 (0 indicating no arthritis and 100 indicating extremely active arthritis); participant's pain assessment using VAS on a scale of 0-100 (0 indicating no pain and 100 indicating severe pain); health assessment questionnaire-disability index (HAQ-DI) score contains 20 questions,8 components: dressing/ grooming, arising, eating, walking, hygiene, reach, grip, and errands/chores and scored on a scale of 0-3 (0 and 3 indicating without difficulty and unable to do); hsCRP.
Percentage of Participants Who Achieve ACR 50% Improvement (ACR50) Response at Week 12 | Week 12
  ACR50 response is achieved when the participant has: ≥ 50% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA assessed using VAS on a scale of 0-100 (0 indicating no disease activity and 100 indicating maximum disease activity) and SGA assessed using VAS on a scale of 0-100 (0 indicating no arthritis and 100 indicating extremely active arthritis); participant's pain assessment using VAS on a scale of 0-100 (0 indicating no pain and 100 indicating severe pain); HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and errands/chores and scored on a scale of 0-3 (0 and 3 indicating without difficulty and unable to do); hsCRP.
Percentage of Participants Who Achieve ACR 70% Improvement (ACR70) Response at Week 12 | Week 12
  ACR70 response is achieved when the participant has: ≥ 70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA assessed using VAS on a scale of 0-100 (0 indicating no disease activity and 100 indicating maximum disease activity) and SGA assessed using VAS on a scale of 0-100 (0 indicating no arthritis and 100 indicating extremely active arthritis); participant's pain assessment using VAS on a scale of 0-100 (0 indicating no pain and 100 indicating severe pain); HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and errands/chores and scored on a scale of 0-3 (0 and 3 indicating without difficulty and unable to do); hsCRP.
Change From Baseline in Simplified Disease Activity Index (SDAI) at Week 12 | Baseline, Week 12
  SDAI is a composite measure that sums the TJC28, SJC28, SGA, PGA, and the hsCRP (in mg/dL). PGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no disease activity and maximum disease activity) and SGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no arthritis and extremely active arthritis). Higher score indicates more severe disease activity status and total possible score is 0 to 86. A negative change from baseline indicates improvement.
Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 12 | Baseline, Week 12
  CDAI is calculated using formula: CDAI = TJC based on 28 joints (TJC28) + SJC based on 28 joints (SJC28) + SGA + PGA. PGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no disease activity and maximum disease activity) and SGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no arthritis and extremely active arthritis). CDAI can range from 0 to 76, with higher score indicating more severe disease activity status. A negative change from baseline indicates improvement.
Percentage of Participants Who Achieve SDAI ≤ 11 at Week 12 | Week 12
  SDAI is a composite measure that sums the TJC28, SJC28, SGA, PGA, and the hsCRP (in mg/dL). PGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no disease activity and maximum disease activity) and SGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no arthritis and extremely active arthritis). Higher score indicates more severe disease activity status and total possible score is 0 to 86.
Percentage of Participants Who Achieve CDAI ≤ 10 at Week 12 | Week 12
  CDAI is calculated using formula: CDAI = TJC based on 28 joints (TJC28) + SJC based on 28 joints (SJC28) + SGA + PGA. PGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no disease activity and maximum disease activity) and SGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no arthritis and extremely active arthritis). CDAI can range from 0 to 76, with higher score indicating more severe disease activity status.
Percentage of Participants Who Achieve DAS28(CRP) ≤ 3.2 at Week 12 | Week 12
  The DAS28(CRP) is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA and hsCRP measurement for a total possible score of 1 to 9.4. Higher values indicate higher disease activity.
Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 12 | Baseline, Week 12
  The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 domains (dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and errands/chores). Responses are scored on a 4-point Likert scale from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. The need for aids or help from another person will also be recorded. The HAQ-DI total score ranges from 0 to 3 with higher scores indicating greater dysfunction. Negative change from baseline indicates improvement (less disability).
Percentage of Participants Who Achieve SDAI ≤ 3.3 at Week 12 | Week 12
  SDAI is a composite measure that sums the TJC28, SJC28, SGA, PGA, and the hsCRP (in mg/dL). PGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no disease activity and maximum disease activity) and SGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no arthritis and extremely active arthritis). Higher score indicates more severe disease activity status and total possible score is 0 to 86.
Percentage of Participants Who Achieve CDAI ≤ 2.8 at Week 12 | Week 12
  CDAI is calculated using formula: CDAI = TJC based on 28 joints (TJC28) + SJC based on 28 joints (SJC28) + SGA + PGA. PGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no disease activity and maximum disease activity) and SGA assessed using VAS on a scale of 0-10 (0 and 10 indicating no arthritis and extremely active arthritis). CDAI can range from 0 to 76, with higher score indicating more severe disease activity status.
Percentage of Participants Who Achieve DAS28(CRP) < 2.6 at Week 12 | Week 12
  The DAS28(CRP) is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA, and hsCRP measurement for a total possible score of 1 to 9.4. Higher values indicate higher disease activity.
Pharmacokinetic (PK) Parameter: AUCtau of GS-5718 | Up to Week 12
  AUCtau is defined as the area under the curve from time zero to end of dosing interval.
PK Parameter: AUCtau of Methotrexate (MTX) | Up to Week 8
  AUCtau is defined as the area under the curve from time zero to end of dosing interval.
PK Parameter: Cmax of GS-5718 | Up to Week 12
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: Cmax of MTX | Up to Week 8
  Cmax is defined as the maximum observed concentration of drug.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-561-5898